CLINICAL TRIAL: NCT00684775
Title: Employment-Based Depot Naltrexone Clinical Trial II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-19497-2; R01DA019497-02 (NIH); NA_00000928 (Other: Johns Hopkins Medicine IRB)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Work Plus Naltrexone Prescription (No Intervention): Participants could work and earn vouchers but did not to take Vivitrol Injections to work and earn vouchers.
- Work Plus Naltrexone Contingency (Experimental): Participants could work and earn vouchers and had to take Vivitrol Injections to work and earn vouchers: employment-based reinforcement.
  Interventions: Combination Product: Work Plus Naltrexone Contingency

INTERVENTIONS:
Combination Product: Work Plus Naltrexone Contingency — Vivitrol, an extended-release depot formulation of naltrexone, was used. Participants were offered an inpatient opioid detoxification and oral naltrexone induction. Participants who complete the oral naltrexone induction (N=40) were randomly assigned to one of two groups. Both groups will be invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone for 6 months. Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections once per month.
  Other Names: contingency management
  Arms: Work Plus Naltrexone Contingency

SUMMARY:
The purpose of this study is to determine whether employment-based naltrexone treatment proves effective in promoting depot naltrexone adherence and drug abstinence.

DETAILED DESCRIPTION:
A randomized study is planned to evaluate the effectiveness of employment-based reinforcement in promoting depot naltrexone adherence in opiate-dependent adults. Vivitrol, an extended-release depot formulation of naltrexone approved by the FDA for the treatment of alcohol dependence, will be used. Participants will be offered an inpatient opioid detoxification and oral naltrexone induction. Participants who complete the oral naltrexone induction (N=40) will be randomly assigned to one of two groups. Both groups will be invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone for 6 months. Participants in the "Work Plus Naltrexone Contingency" condition will earn access to working and earning salary by taking depot naltrexone injections once per month. "Work Plus Naltrexone Prescription" participants will be encouraged to take depot naltrexone monthly, but access to working and earning salary will not be contingent on doing so.

ELIGIBILITY:
Individuals were eligible if they:

* met the Diagnostic and Statistical Manual (DSM)-IV criteria for opioid dependence,
* reported using heroin at least 21 of the last 30 days while living in the community,
* were unemployed,
* were 18-65 years old,
* were medically approved for naltrexone,
* lived in or near Baltimore, MD.

Individuals were excluded if they:

* were pregnant or breastfeeding,
* had serum aminotransferase levels over three times normal,
* had current hallucinations, delusions, or thought disorders, current suicidal or -homicidal ideation,
* expressed interest in methadone treatment,
* were required to use opioids for medical purposes,
* earned over $200 in taxable income over the previous 30 days,
* had physical limitations that would prevent them from using a keyboard, or were incarcerated or under constant monitoring by the criminal justice system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2010-04-30 (Actual); Study Completion 2010-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Professor, Johns Hopkins University School of Medicine
Locations (1):
- The Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] DeFulio A, Everly JJ, Leoutsakos JM, Umbricht A, Fingerhood M, Bigelow GE, Silverman K. Employment-based reinforcement of adherence to an FDA approved extended release formulation of naltrexone in opioid-dependent adults: a randomized controlled trial. Drug Alcohol Depend. 2012 Jan 1;120(1-3):48-54. doi: 10.1016/j.drugalcdep.2011.06.023. Epub 2011 Jul 22. PMID 21782353

RESULTS

PARTICIPANT FLOW:
Groups:
- Work Plus Naltrexone Prescription: Participants who completed the oral naltrexone induction (N=38) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone for 6 months. Participants in the "Work Plus Naltrexone Prescription" condition could work and earn salary independent of whether or not they took depot naltrexone injections.
- Work Plus Naltrexone Contingency: Participants who completed the oral naltrexone induction (N=38) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone for 6 months. "Work Plus Naltrexone Contingency" participants were required to take monthly depot naltrexone injections to work and earn salary.
Period: Overall Study
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 Work Plus Naltrexone Prescription: Work Plus Naltrexone Prescription
  employment-based reinforcement: Vivitrol, an extended-release depot formulation of naltrexone, will be used. Participants will be offered an inpatient opioid detoxification and oral naltrexone induction. Participants who complete the oral naltrexone induction (N=40) will be randomly assigned to one of two groups. Both groups will be invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone for 6 months. Participants in the "Work Plus Naltrexone Contingency" condition will earn access to working and earning salary by taking depot naltrexone injections once per month. "Work Plus Naltrexone Prescription" participants will be encouraged to take depot naltrexone monthly, but access to working and earning salary will not be contingent on doing so.
- 2 Work Plus Naltrexone Contingency: Work Plus Naltrexone Contingency
  employment-based reinforcement: Vivitrol, an extended-release depot formulation of naltrexone, will be used. Participants will be offered an inpatient opioid detoxification and oral naltrexone induction. Participants who complete the oral naltrexone induction (N=40) will be randomly assigned to one of two groups. Both groups will be invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone for 6 months. Participants in the "Work Plus Naltrexone Contingency" condition will earn access to working and earning salary by taking depot naltrexone injections once per month. "Work Plus Naltrexone Prescription" participants will be encouraged to take depot naltrexone monthly, but access to working and earning salary will not be contingent on doing so.
- Total: Total of all reporting groups
Arm/Group | 1 Work Plus Naltrexone Prescription | 2 Work Plus Naltrexone Contingency | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (10) | 45 (8) | 44 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 8 | 14 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 16 | 18 | 34
  White | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Naltrexone Injections Received
Description: The percentage of depot naltrexone doses that participants received
Time Frame: 24 weeks
Population: intent-to-treat
Measure: Mean (Full Range); unit: Percentage of injections received
Groups:
- Work Plus Naltrexone Prescription: Participants who completed the oral naltrexone induction (N=38) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone injections for 6 months. Participants in the "Work Plus Naltrexone Prescription" condition could work and earn wages independent of whether or not the took scheduled injections.
- Work Plus Naltrexone Contingency: Participants who completed the oral naltrexone induction (N=38) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone for 6 months. Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections once per month.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 19 | 19
Percentage of injections received | 51.8 [0 to 100] | 86.8 [33 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.002, General Estimating Equation (GEE); Odds Ratio (OR) = 6.0, 95% CI 2-sided [1.44 to 25.0]

2. Primary Outcome: Time to the First Missed Dose
Description: The time to the first missed dose of depot naltrexone
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Work Plus Naltrexone Prescription: Participants could work and earn vouchers but did not to take naltrexone to work and earn vouchers.
- Work Plus Naltrexone Contingency: Participants could work and earn vouchers and had to take naltrexone to work and earn vouchers: employment-based reinforcement.
  employment-based reinforcement: Vivitrol, an extended-release depot formulation of naltrexone, will be used. Participants will be offered an inpatient opioid detoxification and oral naltrexone induction. Participants who complete the oral naltrexone induction (N=40) will be randomly assigned to one of two groups. Both groups will be invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone for 6 months. Participants in the "Work Plus Naltrexone Contingency" condition will earn access to working and earning salary by taking depot naltrexone injections once per month. "Work Plus Naltrexone Prescription" participants will be encouraged to take depot naltrexone monthly, but access to working and earning salary will not be contingent on doing so.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 19 | 19
weeks | 14.74 (7.67) | 20.84 (5.59)
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.0081, t-test, 2 sided

3. Secondary Outcome: Percentage of 30-day Urine Samples Negative for Opiates
Description: Percentage of urine samples collected at the 30-day assessments that are negative for opiates
Time Frame: Collected every 30 days for 150 days
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of opiate negative
Groups:
- Work Plus Naltrexone Prescription: Participants who completed the oral naltrexone induction (N=38) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone injections for 6 months. Participants in the "Work Plus Naltrexone Prescription" condition could work and earn wages independent of whether or not the took scheduled injections.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 19 | 19
percentage of opiate negative | 65.3 [0 to 100] | 71.6 [0 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.56, General Estimating Equation (GEE); Odds Ratio (OR) = 1.34, 95% CI 2-sided [.5 to 3.6]

4. Secondary Outcome: Percentage of M-W-F Samples Negative for Cocaine
Description: Percentage of urine samples collected Monday, Wednesday and Friday at the workplace that are negative for cocaine
Time Frame: Collected every Monday, Wednesday and Friday for 24 weeks
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of mwf cocaine negative
Groups:
- Work Plus Naltrexone Prescription: Participants who completed the oral naltrexone induction (N=38) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone for 6 months. "Work Plus Naltrexone Prescription" participants were encouraged to take depot naltrexone monthly, but access to working and earning salary was not contingent on doing so.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 19 | 19
percentage of mwf cocaine negative | 45.3 [0 to 97] | 54.6 [1 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.41, General Estimating Equation (GEE); Odds Ratio (OR) = 1.45, 95% CI 2-sided [.6 to 3.53]

5. Secondary Outcome: Average Percentage of 30-day Urine Samples Negative for Cocaine
Description: The percentage of urine samples collected at 30-day assessments that are negative for cocaine.
Time Frame: Collected every 30 days for 150 days
Population: intent to treat
Measure: Mean (Full Range); unit: percentage cocaine negative urine sample
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 19 | 19
percentage cocaine negative urine sample | 53.7 [0 to 100] | 57.9 [0 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.75, General Estimating Equation (GEE); Odds Ratio (OR) = 1.19, 95% CI 2-sided [.42 to 3.36]

6. Secondary Outcome: HIV Risk Behaviors
Description: behaviors that place participants at risk for acquiring or transmitting HIV infection
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of months reported
Groups:
- Work Plus Naltrexone Prescription: Participants who complete the oral naltrexone induction (N=38)were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone for 6 months."Work Plus Naltrexone Prescription" participants were encouraged to take depot naltrexone monthly, but access to working and earning salary was not contingent on doing so.
- Work Plus Naltrexone Contingency: Participants who complete the oral naltrexone induction (N=38) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone for 6 months. Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections once per month.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 19 | 19
percentage of months reported | 2.1 (14.4) | 0 (0)
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.1543, t-test, 2 sided

7. Secondary Outcome: Percentage of M,W,F Urine Samples Negative for Opiates
Description: Percentage of urine samples collected Monday, Wednesday and Friday at the workplace that are negative for opiates
Time Frame: Collected every Monday, Wednesday and Friday for 24 weeks
Population: intent to treatment
Measure: Mean (Full Range); unit: percentage of opiate negative
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 19 | 19
percentage of opiate negative | 51.8 [4 to 99] | 66.2 [7 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.15, General Estimating Equation (GEE); Odds Ratio (OR) = 1.82, 95% CI 2-sided [.81 to 4.1]

ADVERSE EVENTS:
Time Frame: Every month for 6 months
Arm/Group | 1 Work Plus Naltrexone Prescription | 2 Work Plus Naltrexone Contingency
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 2/19 | 4/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Work Plus Naltrexone Prescription (N=19) | 2 Work Plus Naltrexone Contingency (N=19)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Reduced sex drive (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sleeplessness (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No